CLINICAL TRIAL: NCT05730959
Title: Sacral Nerve Modulation in IPAA Patients With Poor Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Tom Oresland, Clinical professor, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/2206
Record Dates: First submitted 2019-04-30; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Stoma Malfunction
Keywords: IPAA (Ileal Pouch-Anal Anastomosis); SNM (Sacral Nerve Modultion)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- malfunctioning IPAA (Other): Patients with malfunctioning IPAA
  Interventions: Device: Sacral nerve modulation

INTERVENTIONS:
Device: Sacral nerve modulation — Implant of nerve stimulator

SUMMARY:
IPAA patients with poor functional outcome where no obvious reason can be detected are identified from our patient registry. These patients are offered a sacral nerve modulation test period of three weeks. They will then be scored on function and physiological testing will be done by a Barostat. After a another 14 days without stimulation the tests will be repeated. Those who respond positively will be offered permanent implantation of the Device..

ELIGIBILITY:
Inclusion Criteria:

* UC With IPAA
* Bad functional outcome

Exclusion Criteria:

* Established treatable cause of malfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Øresland Score | 12 months
  functional score

SECONDARY OUTCOMES:
Bowel physiology | At inclusion and at 12 months
  Barostat

CONTACTS AND LOCATIONS:
Overall Officials: Tom Oresland, PhD, Study Chair — University of Oslo

IPD SHARING:
Plan to Share IPD: No